CLINICAL TRIAL: NCT06863038
Title: Predictive Value of the PREMM5, MMRpredict Models, and the Universal Tumor Screening Strategy for Lynch Syndrome in Vietnam
Brief Title: Predictive Value of PREMM5, MMRpredict, and Universal Tumor Screening for Lynch Syndrome in Vietnam
Acronym: Predict_LS_VN
Status: Not yet recruiting | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: Gene Solutions (Industry)
Responsible Party: Principal Investigator, Doan Thi Nha Nguyen, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: VN_Predict_Lynch_241223
Record Dates: First submitted 2025-02-28; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Lynch Syndrome; Colorectal Cancer (CRC)
Keywords: Lynch Syndrome; Universal Tumor Screening; Colorectal cancer; PREMM5; MMRpredict
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — This study will retain formalin-fixed paraffin-embedded (FFPE) tumor tissue samples and peripheral blood samples collected from participants.
  Tumor biopsy specimens will be obtained during colonoscopy and used for histopathological analysis, immunohistochemistry (IHC), BRAF V600E mutation analysis, and MLH1 methylation assessment.
  Blood samples (2 mL in EDTA tubes) will be used for germline DNA extraction and Next-Generation Sequencing (NGS) for MMR gene mutations.
  Tumor tissue may also undergo somatic MMR gene sequencing in cases without germline mutations. Samples will be stored securely at -80°C for blood DNA and at room temperature for FFPE blocks following institutional biorepository guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study evaluates the predictive value of PREMM5, MMRpredict models, and Universal Tumor Screening in detecting Lynch Syndrome in colorectal cancer (CRC) patients in Vietnam.

Vietnamese CRC patients (18-70 years) undergoing colonoscopy will be enrolled. Participants will complete a medical history questionnaire and provide blood samples for genetic testing. Tumor biopsy specimens will undergo Immunohistochemistry staining, BRAF V600E mutation, and MLH1 methylation analysis in case of loss of MLH1/PMS2 expression. Next-Generation Sequencing will detect germline MMR mutations, and biallelic somatic mutations will be analyzed if no germline mutations are found.

DETAILED DESCRIPTION:
1. Background and Rationale Colorectal cancer (CRC) is one of the most prevalent malignancies worldwide and the second leading cause of cancer-related deaths. Approximately 5-6% of CRC cases are associated with hereditary cancer syndromes, with Lynch Syndrome (LS) being the most common. LS results from germline mutations in the Mismatch Repair (MMR) genes (MLH1, MSH2, MSH6, PMS2, and EPCAM), which lead to microsatellite instability (MSI) and an increased risk of CRC, endometrial, and other extracolonic malignancies.

   Despite its significance, LS remains underdiagnosed, particularly in Asian populations, due to the limitations of traditional screening criteria, such as Amsterdam II and the Revised Bethesda Guidelines, which have low sensitivity in identifying LS patients. In response, universal tumor-based screening using MSI testing and immunohistochemistry (IHC) for MMR protein loss has been proposed as an effective alternative. Additionally, prediction models such as PREMM5 and MMRpredict have been developed to estimate LS risk based on clinical and family history.

   However, these models and tumor screening strategies have not been validated in the Vietnamese population. This study aims to evaluate and compare the predictive performance of different screening approaches for LS in Vietnamese CRC patients, thereby optimizing genetic testing selection and early diagnosis.
2. Study Design and Setting

   This is a cross-sectional study conducted at two major hospitals in Vietnam:
   * University Medical Center at Ho Chi Minh City - GI Endoscopy Department
   * Nguyen Tri Phuong Hospital - GI Endoscopy & Gastrointestinal Surgery Departments The study will enroll CRC patients aged 18-70 years who undergo colonoscopy with suspected tumors and are subsequently diagnosed with colorectal adenocarcinoma.
3. Objectives

   Primary Objective:

   - To assess the predictive value of PREMM5, MMRpredict, and Universal Tumor Screening Strategy in detecting Lynch Syndrome in CRC patients.

   Secondary Objectives:
   * To determine the prevalence of Lynch Syndrome based on germline MMR gene mutation testing.
   * To describe the clinical characteristics of Lynch Syndrome-Associated CRCs.
   * To describe the the endoscopic and histopathological features of Lynch Syndrome-Associated CRCs
   * To compare the diagnostic accuracy (AUC-ROC, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV)) of different screening models and criteria, including Amsterdam II, Revised Bethesda Guidelines, PREMM5, MMRpredict, and Universal Tumor Screening.
4. Study Procedures Patient Enrollment & Sample Collection

   Eligible patients will:
   * Provide informed consent before participation.
   * Complete a medical history questionnaire assessing:

     * Family history of CRC and LS-related cancers.
     * Personal history of CRC, endometrial, and other extracolonic malignancies.
     * Clinical symptoms and lifestyle risk factors.
   * Provide a 2 mL blood sample for germline genetic testing.
5. Laboratory Analysis

   * Histopathological Evaluation: Tumor biopsy samples will be fixed in formalin, sectioned, and stained for Hematoxylin-Eosin (H&E) evaluation.
   * MMR Protein Expression: IHC will assess the loss of MLH1, MSH2, MSH6, and PMS2 expression.
   * BRAF V600E Mutation & MLH1 Methylation: Tumors with MLH1/PMS2 loss will undergo further testing to determine sporadic vs. hereditary LS cases.
   * Germline MMR Mutation Testing: All the blood samples will undergo Next-Generation Sequencing (NGS) to detect pathogenic germline MMR mutations.
   * Biallelic Somatic Mutation Analysis: If no germline mutations are identified in case of MLH1/PMS2 expression loss and no BRAF V600E mutation and no MLH1 methylation, tumor tissue sequencing will determine biallelic somatic inactivation.
6. Statistical Considerations Sample Size Calculation The sample size is calculated based on the estimated prevalence of LS at 2.9%, requiring at least 572 participants (including a 10% dropout rate) to achieve statistical power.
7. Statistical Analysis

   * Quantitative variables (e.g., age, tumor size) will be expressed as mean ± standard deviation or median with interquartile range.
   * Categorical variables (e.g., IHC results, BRAF V600E mutation) will be reported as percentages.
   * Diagnostic performance will be evaluated using Receiver Operating Characteristic (ROC) curves, sensitivity, specificity, PPV, and NPV.
   * Comparison of screening models (Amsterdam II, Bethesda, PREMM5, MMRpredict, Universal Tumor Screening) will be based on their AUC-ROC values.
   * Significance level: p < 0.05.
8. Ethical Considerations This study adheres to Good Clinical Practice (GCP) and the Declaration of Helsinki. Ethical approval has been obtained from the Institutional Review Board (IRB), and all participants will provide written informed consent.

   * Patient confidentiality will be ensured by de-identifying all study data.
   * All data will be retained for at least three years post-study completion. Data Quality and Monitoring
   * Standard Operating Procedures (SOPs): Guidelines will be followed for sample collection, DNA extraction, MSI/IHC testing, and genetic analysis.
   * Plan for Missing Data: Cases with missing or inconsistent data will be reviewed, and statistical methods such as multiple imputation will be used if necessary.
   * Registry Oversight & Compliance: The study will follow national biomedical research regulations and ensure compliance with international registry requirements (e.g., ClinicalTrials.gov).
9. Study Duration and Expected Outcomes

   - Study Duration: 24 months (March 2025 - March 2027).
10. Expected Outcomes:

    * Improved LS detection rates in Vietnamese CRC patients.
    * Validation of prediction models (PREMM5, MMRpredict) in the Vietnamese population.
    * Enhanced cost-effectiveness in LS screening and genetic testing selection.
    * Contribution to national screening guidelines for hereditary cancer syndromes. By refining LS screening strategies, this study will support early cancer detection, preventive interventions, and genetic counseling in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years
* Provide informed consent to participate in the study
* Undergo colonoscopy with endoscopic findings suspicious for CRC
* Have biopsy-confirmed adenocarcinoma through colonoscopic biopsy

Exclusion Criteria:

* Active gastrointestinal bleeding
* Currently using anticoagulants or antiplatelet agents
* History of coagulation disorders or difficulty controlling bleeding
* Incomplete colonoscopy to the cecum (excluding cases of tumor-induced obstruction)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include Vietnamese patients aged 18-70 years who undergo colonoscopy at the University Medical Center Ho Chi Minh City and Nguyen Tri Phuong Hospital with suspected colorectal tumors. Eligible participants will be those diagnosed with colorectal adenocarcinoma through biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of PREMM5, MMRpredict, and Universal Tumor Screening for Lynch Syndrome in Colorectal Cancer Patients | At study completion (Month 24). The primary outcome will be analyzed after all participants have completed sample collection, genetic testing, and data processing, expected within 24 months from study initiation.
  The study evaluates the diagnostic accuracy of PREMM5, MMRpredict models, and Universal Tumor Screening (IHC testing) in detecting Lynch Syndrome (LS) in colorectal cancer (CRC) patients. The outcome will be assessed by calculating sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the receiver operating characteristic curve (AUC-ROC) for each screening method compared to gold-standard germline MMR gene mutation testing (via Next-Generation Sequencing - NGS).

SECONDARY OUTCOMES:
Prevalence of Lynch Syndrome in Colorectal Cancer Patients | At study completion (Month 24)
  This outcome measures the proportion of colorectal cancer (CRC) patients diagnosed with Lynch Syndrome (LS) based on germline MMR gene mutation testing (via Next-Generation Sequencing - NGS). The prevalence will be reported as a percentage of the total study population.
Clinical Characteristics of Lynch Syndrome-Associated CRC | At study completion (Month 24)
  This outcome describes the clinical characteristics of Lynch Syndrome-associated CRC vs. sporadic CRC. Key characteristics include age at CRC diagnosis, personal history of cancer and age of onset, family history of cancer and age at diagnosis, and clinical symptoms.
Endoscopic and histopathological features of Lynch Syndrome-Associated CRC | At study completion (Month 24)
  This outcome describes the endoscopic and histopathological features of Lynch Syndrome vs. sporadic CRC tumors. Key characteristics include tumor location, tumor quantity, and histopathological features.
Comparison of Screening Criteria and Prediction Models for Lynch Syndrome | At study completion (Month 24)
  This outcome compares the diagnostic accuracy (sensitivity, specificity, PPV, NPV, and AUC-ROC) of different LS screening methods, including Amsterdam II Criteria, Revised Bethesda Guidelines, PREMM5 Model, MMRpredict Model, and Universal Tumor Screening (IHC testing).

CONTACTS AND LOCATIONS:
Overall Officials: Doan TN Nguyen, MD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No